CLINICAL TRIAL: NCT02996084
Title: Longitudinal Brain Volume Change (and Correlates) in Healthy Control Subjects: A Normative Sub-Study of Multiple Sclerosis Partners Advancing Technology and Health Solutions (MS PATHS)
Brief Title: MS PATHS Normative Sub-Study
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 888MS005
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteer
Keywords: Imaging research

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ribonucleic acid (RNA), serum, and whole blood biomarker samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this study is to determine the normative range of brain volume and brain volume change in healthy control (HC) participants whose age, race, and gender distribution is approximately matched to the age, race, and gender distribution of patients with Multiple Sclerosis (MS) enrolled in Study 888MS001. The secondary objective is to use the results of the primary endpoint to ensure consistency of brain volume measurements across MS PATHS centers.

ELIGIBILITY:
Key Inclusion Criteria

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local participant privacy regulations.

Key Exclusion Criteria

* History of human immunodeficiency virus.
* Confirmed or suspected pregnancy.
* Diagnosis of migraine requiring medication or any other participant-reported diagnosis of a neurological disease or condition (e.g., stroke, transient ischemic attack, epilepsy, brain infection, brain surgery, prior head injury or concussion, or brain tumor).
* Any participant-reported diagnosis of an autoimmune disorder (e.g., rheumatoid arthritis, Sjögren's syndrome, scleroderma, or systemic lupus erythematosus).
* Standard MRI exclusion criteria, including claustrophobia, inability to lay still in the magnet (e.g., tremor), or any type of implanted metal in the body that would be affected by the strong magnetic field.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy control (HC) participants enrolled at each institution will be carefully selected to result in a group whose age, race, and gender distribution is approximately matched to the age, race, and gender distribution of patients with MS enrolled in MS PATHS at that center. Patients enrolled in MS PATHS at each center will be encouraged to enlist a friend or family member to participate in the study as an HC. Subsequently, on approximately quarterly review of participant participation, particular demographic groups will be targeted for recruitment, if needed, in order for the age, race, and gender distribution of a center's HC sample to be similar to their MS PATHS participant sample (within the study age range).
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Brain volume | Every 12 months up to 3 years
  Measured by using magnetic resonance imaging (MRI) scans
Brain volume change | Every 12 months up to 3 years
  Measured by using MRI scans

SECONDARY OUTCOMES:
Development of models to calibrate brain volume measurements between centers, if necessary | Up to 3 years
  Measured by using MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (6):
- United States (4):
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
- University Hospital Carl Gustav Carus Dresden, Dresden, Germany
- Multiple Sclerosis Centre of Catalonia (Cemcat) Vall d'Hebron Hospital, Barcelona, Spain